CLINICAL TRIAL: NCT00544778
Title: Phase II Trial of Neoadjuvant Dose-Dense Doxorubicin, Ifosfamide, and Irinotecan (CPT-11) for Advanced Soft Tissue and Recurrent Bone Sarcomas
Brief Title: Combination Chemotherapy and Dexrazoxane Followed by Surgery and Radiation Therapy in Treating Patients With Advanced Soft Tissue Sarcoma or Recurrent Bone Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely due to withdrawal of support by the sponsor.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00050; P30CA033572 (NIH); CHNMC-00050; CDR0000566381 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; metastatic osteosarcoma; recurrent osteosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; Ewing sarcoma of bone
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Filgrastim; Dexrazoxane; Doxorubicin; Ifosfamide; Irinotecan; Immunoenzyme Techniques; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

ARMS (1):
- Arm 1 (Experimental): High-dose chemotherapy with doxorubicin at 120 mg/m2 and ifosfamide at 2 g/m2 followed by a prolonged schedule of CPT-11 at 20 mg/m2.
  Interventions: Biological: filgrastim; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: ifosfamide; Drug: irinotecan hydrochloride; Genetic: protein expression analysis; Other: immunoenzyme technique; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: dexrazoxane hydrochloride
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: irinotecan hydrochloride
Genetic: protein expression analysis
Other: immunoenzyme technique
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin, ifosfamide, and irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Chemoprotective drugs, such as dexrazoxane, may protect normal cells from the side effects of chemotherapy. Giving combination chemotherapy together with dexrazoxane before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with dexrazoxane followed by surgery and radiation therapy works in treating patients with advanced soft tissue sarcoma or recurrent bone sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the effectiveness of neoadjuvant dose-dense chemotherapy comprising doxorubicin hydrochloride, ifosfamide, and irinotecan hydrochloride in combination with dexrazoxane hydrochloride followed by surgery and radiotherapy in patients with advanced soft tissue sarcoma or recurrent bone sarcoma.
* To evaluate the toxicities of this regimen in these patients.
* To compare the duration of disease-free and overall survival of patients with advanced soft tissue sarcoma who receive this therapy on a neoadjuvant basis with historical controls.
* To evaluate laboratory correlates of chemotherapy resistance for the cytotoxic agents used in this study.

OUTLINE: Patients are stratified by type of sarcoma (soft tissue vs bone), prior treatment (untreated vs treated), and presence of metastases (yes vs no).

* Courses 1 and 2: Patients receive doxorubicin hydrochloride and dexrazoxane hydrochloride IV continuously over 96 hours. Treatment repeats every 3 weeks for 2 courses.
* Courses 3 and 4: Patients receive ifosfamide IV over 2 hours twice a day (every 12 hours) on days 1-3. Treatment repeats every 3 weeks for 2 courses.
* Courses 5 and 6: Patients receive irinotecan hydrochloride IV over 1 hour once a day on days 1-5 and 8-12. Treatment repeats every 3 weeks for 2 courses.

Patients also receive filgrastim (G-CSF) subcutaneously once a day beginning 3 days after completion of chemotherapy and continuing until blood counts recover.

Patients then undergo standard surgery and radiotherapy.

Patients undergo blood sample collection periodically for correlative studies. Samples are analyzed for MDR (multidrug resistance gene) protein expression via immunoperoxidase staining.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 2 years, and then once a year thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Primary soft tissue sarcoma at high-risk* for recurrence, meeting any of the following criteria:

    * Previously untreated locally advanced, nonmetastatic disease
    * Advanced (metastatic) disease not amenable to standard or higher priority investigational neoadjuvant therapies
  * Recurrent bone sarcoma (e.g., osteogenic sarcoma, Ewing sarcoma, or peripheral neuroectodermal tumor)

    * Must have advanced locally recurrent or metastatic disease NOTE: *High-risk is defined as high-grade, deep to fascia, and > 5 cm in greatest dimension
* Measurable or nonmeasurable disease is not required
* Pre-chemotherapy consultation with surgery and radiation oncology is required for formulation of loco-regional therapy
* No gastrointestinal stromal cell sarcoma
* No alveolar soft part sarcoma
* No symptomatic brain metastases

  * No requirement for anticonvulsant or corticosteroid therapy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 2 months
* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count > 120,000/mm^3
* Creatinine clearance > 50 mL/min
* Serum bilirubin ≤ 1.5 mg/dL
* SGOT or SGPT ≤ 2.5 times upper limit of normal
* Serum albumin ≥ 2.5 mg/dL
* LVEF ≥ 50% by MUGA scan
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No concurrent nonmalignant illness (e.g., cardiovascular, pulmonary, or CNS disease) that is poorly controlled with currently available treatment or is of such severity that the investigators deem it unwise for the patient to enter the study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for recurrent (local or metastatic) soft tissue sarcoma
* Prior chemotherapy for recurrent bone sarcoma allowed provided the total dose of doxorubicin hydrochloride is ≤ 300 mg/m^2
* No prior radiotherapy to > 25% of bone marrow
* At least 3 weeks since prior radiotherapy or chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-08; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren A. Chow, MD, Study Chair — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 39 [20 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate defined as the proportion of subjects with confirmed partial or complete response as defined by the RECIST criteria.
Time Frame: First disease evaluation one month after the start of treatment and every 3 months there after, up to 2 years.
Measure: Number; unit: percentage of patients responding
Arm/Group | Arm 1
Number analyzed (Participants) | 7
percentage of patients responding | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 11 months.
Description: "Other" adverse events are all grades and attributions to treatment not included in "Serious" adverse events.
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (21)
Packed red blood cell transfusion (Blood and lymphatic system disorders) | 3 (5)
Sinus tachycardia (Cardiac disorders) | 3 (5)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Incontinence NOS (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (17)
Vomiting (Gastrointestinal disorders) | 6 (11)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 2 (2)
Fatigue (General disorders) | 6 (22)
Fever (General disorders) | 1 (1)
Oedema NOS (General disorders) | 2 (2)
Pain (General disorders) | 4 (8)
Catheter related infection (Infections and infestations) | 1 (1)
Infection NOS (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4)
Alkaline phosphatase increased (Investigations) | 4 (9)
Aspartate aminotransferase increased (Investigations) | 5 (12)
Creatinine increased (Investigations) | 2 (2)
Hyperbilirubinemia (Investigations) | 2 (2)
INR increased (Investigations) | 1 (1)
Leukopenia (Investigations) | 2 (4)
Lymphopenia (Investigations) | 3 (8)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (3)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (11)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (9)
Hypokalemia (Metabolism and nutrition disorders) | 5 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 6 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Depressed level of consciousness (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 6 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (6)
Anxiety (Psychiatric disorders) | 2 (3)
Confusion (Psychiatric disorders) | 3 (5)
Depression (Psychiatric disorders) | 2 (2)
Hallucination NOS (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (5)

LIMITATIONS AND CAVEATS:
The study was terminated…protocol objectives not met. It was closed prematurely due to withdrawal of support by the sponsor. Subjects have been followed, but there is not enough data generated to continue following the subjects."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes